CLINICAL TRIAL: NCT07352670
Title: 5 Verbs for Couples: Program Study
Brief Title: 5 Verbs for Couples - Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Allen Barton, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23761
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Relationships, Marital
MeSH Terms: interventions — Family Characteristics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): 5 verbs for couples participants
  Interventions: Behavioral: 5 Verbs for Couples
- Control (No Intervention): No intervention. Waitlist control group

INTERVENTIONS:
Behavioral: 5 Verbs for Couples — The program consists of an overview and three accompanying sessions, each approximately 30-45 minutes in length. The new program developed by the project PI is organized around five verbs to help strengthen couple relationship. For each of the three sessions, content includes information on increasing gratitude between partners, building friendship and connection, addressing challenges and hardships, being a team, communication, and dedication. This psychoeducational program is largely informative in nature, with recommended thought and/or written exercises for individuals to complete regarding how program material applies to their relationship. Individuals are provided a link to access the program and then watch/click through session activities at a time and location of their choosing (similar to an online self-directed training or course).
  Arms: Treatment

SUMMARY:
The current research is designed to implement and evaluate 5 Verbs for Couples, a new relationship education program that can be completed individually or by both partners together. Involvement will entail completing 3 surveys over a 2-month period. After completing the first survey, a subset of individuals will be randomly assigned to participate in a 3-session online program and answer questions about their experience in the program. The remaining individuals will receive access to the program approximately 2 months later, after completing the third survey.

ELIGIBILITY:
Inclusion Criteria:

* A resident of United States
* 18 years of age or older
* Married, engaged, or living with your partner for at least 6 months
* Willing to participate in online relationship-focused programming

Exclusion Criteria:

* Severe form(s) of intimate partner violence are occurring in the relationship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Relationship Satisfaction | Baseline, 1 month follow-up, 2-month follow-up
  Couple satisfaction index
Change in intervention-targeted behavior | Baseline, 1-month follow-up, 2-month follow-up
  5 Verbs for Couples cognitive-behavioral indicators (new measure created for this study)

SECONDARY OUTCOMES:
Change in psychological distress | Baseline, 1-month, 2-month follow-up
  Kessler 6 item psychological distress

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.publish.illinois.edu/fiveverbs/couples